CLINICAL TRIAL: NCT00941720
Title: A Study of Outcomes and Toxicity of Busulfex as Part of a High Dose Chemotherapy Preparative Regimen in Autologous Hematopoietic Stem Cell Transplantation for Patients With Plasma Cell Myeloma
Brief Title: Busulfan, Cyclophosphamide, and Autologous Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1A07
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Busulfan Treatment (Experimental)
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Procedure: autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: busulfan — IV busulfan 0.8 mg/kg every 6 hours x 16 doses
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon; Myelosan
Drug: cyclophosphamide — IV cyclophosphamide 60 mg/kg over 4 hours x 2 days
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Procedure: autologous hematopoietic stem cell transplantation — infusion of autologous hematopoietic stem cells of at least 2.0 x 106 CD34+ cells/kg on day 0

SUMMARY:
RATIONALE: Giving high-dose chemotherapy before an autologous stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. An autologous stem cell transplant may be able to replace the blood-forming cells that were destroyed by the chemotherapy.

PURPOSE: This phase II trial is studying how well giving busulfan together with cyclophosphamide followed by an autologous stem cell transplant works in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare relapse-free survival and overall survival of patients with multiple myeloma treated with IV busulfan vs historical control patients treated with oral busulfan when administered with cyclophosphamide as a conditioning regimen prior to autologous hematopoietic stem cell transplantation.

Secondary

* To compare pulmonary toxicity rates of IV busulfan vs oral busulfan when administered with cyclophosphamide as a conditioning regimen prior to autologous hematopoietic stem cell transplantation.

OUTLINE: Patients receive high-dose busulfan IV every 6 hours on days -8 to -4 and high-dose cyclophosphamide IV over 4 hours on days -3 and -2. Patients undergo autologous hematopoietic stem cell transplantation on day 0.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with a diagnosis of plasma cell myeloma
* Patients with cardiac ejection fraction >= 45% or clearance by Cleveland Clinic Faculty (CCF) cardiologist
* Patients with diffusion capacity of carbon monoxide (DLCO) >= 45% predicted or clearance by CCF pulmonologist
* Patient with previously harvested peripheral blood progenitor cells with a minimum of 2 x 10^6 CD 34+ cells/kg harvested

EXCLUSION CRITERIA:

* Patients receiving total body irradiation
* Non-myeloablative/reduced-intensity conditioning
* Pregnant and breast feeding patients
* Human immunodeficiency virus (HIV) positive
* Patients with serum creatinine > 2.0
* Prior Hematopoietic Stem Cell (HSC) transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-06-11 (Actual); Primary Completion 2013-02-28 (Actual); Study Completion 2013-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. Sobecks, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Busulfan Treatment
Started | 71
Completed | 57
Not Completed | 14
Not completed — Withdrawal by Subject | 1
Not completed — Insurance denied participation | 11
Not completed — ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Busulfan Treatment
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival
Description: Number of participants without progressive disease at the end of the study period, using the definitions for complete response, partial response and progressive disease from the International Myeloma Working Group .
Time Frame: at 6 months
Measure: Number; unit: participants
Arm/Group | Busulfan Treatment
Number analyzed (Participants) | 57
participants | 48

2. Primary Outcome: Overall Survival
Description: Number of patients alive at the end of the study period
Time Frame: at 6 months
Measure: Number; unit: participants
Arm/Group | Busulfan Treatment
Number analyzed (Participants) | 57
participants | 53

3. Secondary Outcome: Pulmonary Toxicity
Description: Toxicity criteria will be assessed and graded according to the National Cancer Institute (NCI) Common Terminology Criteria (CTC) v3.0. Estimated using exact 95% binomial confidence intervals.
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Busulfan Treatment
Number analyzed (Participants) | 57
percentage of participants | 3.5 [0.4 to 12.1]

ADVERSE EVENTS:
Time Frame: 100 days after off treatment
Arm/Group | Busulfan Treatment
Serious Adverse Events (participants affected / at risk) | 12/57
Other Adverse Events (participants affected / at risk) | 5/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan Treatment (N=57)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic reaction - Angioedemia due to ACE Inhibitors (Immune system disorders) | 1 (1)
Blood and lymphatic system disorders - other (Relapsed disease) (Blood and lymphatic system disorders) | 1 (2)
Death NOS (General disorders) | 5 (5)
Dyspenia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Injury, poisoning and procedural complications - Other (patient fell and hit head. Never recovered) (Injury, poisoning and procedural complications) | 1 (2)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Lung Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan Treatment (N=57)
Catheter related infection (Infections and infestations) | 1 (1)
Colitis - diverticulitis (Gastrointestinal disorders) | 1 (1)
Dyspenia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (3)
Gastrointestinal disorders - Clostridium difficile in urine and diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No